CLINICAL TRIAL: NCT02746341
Title: An Observational, Prospective, Multi-center, Natural History Study of Patients With Mucopolysaccharidosis Type IIIA (MPS IIIA)
Brief Title: Natural History Study of Patients With MPS IIIA
Status: Completed | Type: Observational
Sponsor: LYSOGENE (Industry)
Responsible Party: Sponsor
Other Study IDs: P3-LYS-SAF
Record Dates: First submitted 2016-04-15; First posted 2016-04-21 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Mucopolysaccharidosis IIIA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebral Spinal Fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate the clinical progression in patients with MPS IIIA who are untreated with any investigational product and to obtain standardized assessments: neurocognitive, behavioral, sleep-wake habits and effect of MPS IIIA on the quality of life of patients and their families.

DETAILED DESCRIPTION:
This is a multicenter, multinational, longitudinal, observational study in children aged up to and including 9 years, who have been diagnosed with MPS IIIA. The study will detail the natural course of MPS IIIA via standardized clinical, biochemical, neurocognitive, developmental, behavioral and imaging measures. This information is anticipated to inform the design and interpretation of future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Documented MPS IIIA diagnosis
* Children up to and including 9 years of age
* The patient is sufficiently able, in the opinion of the Investigator, to adhere to the study visit schedule and other protocol requirements
* The patient's parent(s) or legal guardian(s) has signed written informed consent, according to the local regulations and after all relevant aspects of the -study have been explained and discussed

Exclusion Criteria:

* The patient is participating in a clinical trial of any potential disease-modifying investigational medicinal product or taking high dose (>100 mg/kg/day) synthetic genistein (patients on low dose or naturally derived genistein can be included in this study).
* The patient has received a hematopoietic stem cell or bone marrow transplant or gene therapy.
* The patient has received enzyme replacement therapy in the last 6 months.
* Homozygous or compound heterozygous for the S298P mutation or the investigator and/or trial steering committee considers the patient not to have the classical severe form of MPS IIIA.
* Individuals with rare and unrelated serious comorbidities e.g. Down syndrome, intraventricular hemorrhage in the new-born period, or extreme low birth weight (<1500 grams).
* Visual or hearing impairment sufficient, in the clinical judgment of the investigator, to preclude cooperation with neurodevelopmental testing. Use of hearing aids is permitted.

Ages: 0 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects diagnosed with MPS IIIA
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
The change from baseline in cognitive function using the Bayley scales of infant and toddler development third edition | Baseline, and every 6 months, for up to 24 months

SECONDARY OUTCOMES:
Change from baseline in the adaptive behavior composite standard score as measured by the Vineland Adaptive Behavior scale | Baseline and every 6 months up to 24 months
Sleep disturbances measured by Actigraphy | Baseline and every 3 months up to 24 months
Patient Quality of Life Questionnaires | Baseline and every 6 months up to 24 months
Change from baseline in total cortical grey matter volume | Baseline, 12 months, 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil
- Armand Trousseau Public Hospital, Paris, France
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Academic Medical Center, Emma Children's Hospital, Amsterdam, Netherlands
- Great Ormond Street Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided